CLINICAL TRIAL: NCT04780191
Title: Investigation of Treatment Using the MyoRegulator® Device in Patients With Spasticity in the Lower Limb Due to Stroke
Acronym: SPAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: PathMaker Neurosystems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C16-124; 2017-A02060-53 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-07-13; First posted 2021-03-03 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Muscle Spasticity; Stroke
Keywords: stroke rehabilitation; spasticity; neuromodulation; trans-spinal direct current stimulation
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active MyoRegulator® treatment (Experimental): Five consecutive days of 20 minutes active stimulation with MyoRegulator® device
  Interventions: Device: MyoRegulator®
- Sham MyoRegulator® treatment (Sham Comparator): Five consecutive days of 20 minutes sham stimulation with MyoRegulator® device
  Interventions: Device: MyoRegulator®

INTERVENTIONS:
Device: MyoRegulator® — Trans-spinal DC stimulation paired with peripheral DC stimulation

SUMMARY:
This is a single center, randomized, double-blind (patient and evaluator), sham-controlled study. The main objectives of this study are to evaluate the performance and safety of the MyoRegulator® device in active versus sham treated stroke patients with lower-limb spasticity after 5 consecutive days of treatment.

DETAILED DESCRIPTION:
Spasticity prevalence after stroke is highly variable, ranging from 17% to 43% three months post-stroke. In the lower limbs, adduction and extension of the knee with equinovarus foot is the most observed pattern. Spasticity can lead to pain, ankylosis, and tendon retraction which may limit the potential success of rehabilitation. Spasticity can also affect quality-of-life and can be highly detrimental to daily activities such as walking.

An initial clinical trial of safety and feasibility suggested that five sessions of treatment with the MyoRegulator® device temporarily reduces spasticity and overall stiffness of the affected extremity with optimal reductions in spasticity occurring 2-3 weeks post stimulation intervention.

MyoRegulator® is a non-invasive neuromodulation device using multi-site direct current stimulation for the treatment of spasticity. The main objectives of this study are to evaluate the performance and safety of the MyoRegulator® device in active versus sham treated patients during and after 5 consecutive days of treatment sessions. Patients can take part in an optional 3-month follow-up.

The primary performance endpoint is defined as the reduction in ankle joint spasticity. The study will be considered to have a successful outcome if the actively treated subjects demonstrate a statistically greater reduction in spasticity, as measured by the Tardieu Scale, as compared to the sham treated subjects after five treatment sessions.

The primary safety endpoint is defined as the incidence of device-related serious adverse events. The safety of the device will be demonstrated if there are no incidents of serious adverse events caused or contributed to by the device treatment that are clinically unacceptable in light of the treatment benefits.

ELIGIBILITY:
Inclusion Criteria:

* Stroke, with cortical and/or subcortical lesions, of at least 6-months duration at study inclusion
* Spasticity in the lower extremity plantarflexors (gastrocnemius, soleus muscles) due to stroke with a baseline score of 1-4 as assessed by the Tardieu scale
* Minimum 1-month duration of spasticity as confirmed by medical history
* Modified Rankin score < 4
* Cognitive functions sufficient to understand the experiments and follow instructions and ability to provide informed consent in accordance with ICH and GCP
* Affiliated with the French social security scheme, universal medical coverages (CMU), or an equivalent scheme.

Exclusion Criteria:

* Enrollment in another biomedical research study at the time of the MyoRegulator study.
* Fixed contractures or profound muscle atrophy in the spastic limb
* Ongoing use of digitalis, morphine, intrathecal pump
* Plantar orthosis or history of orthopedic surgery that can interfere with gait analysis
* Botulinum toxin treatment within 12 weeks of study enrollment
* Prior phenol or alcohol injections within 6 months of study enrollment
* Change in the antispastic treatment (baclofen, clonidine, benzodiazepine, dantrolene, gabapentine, tizanidin) in the 2 months prior to visit 1.
* Allergy to latex
* Presence of potential tsDCS risk factors:

  * Damaged skin at the stimulation sites (i.e., skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, cancerous lesions, etc.)
  * Lack of sensory perception at the stimulation sites
  * Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker, epidural stimulation electrodes, etc.), an intravascular clip or any other electrically sensitive support system
  * Metal in or on the body in the direct path of the stimulation current (jewelry must be removed during stimulation)
  * Past history of seizures or unexplained spells of loss of consciousness during the previous 36 months
* Prior trans-spinal direct current stimulation for any reason or prior trans-cranial direct current stimulation in the past 12 months
* Any medical condition that would prevent the subject from being able to participate in the clinical outcome measures
* Pregnancy in women (as determined by a urine pregnancy test in pre-menopausal women), or lactating women or women planning pregnancy during the course of the study
* Patient under guardianship or curatorship, or under judicial supervision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Change in spasticity from baseline to after the last treatment session | Immediately after last treatment session
  Change in spasticity as measured by the Modified Tardieu Scale (MTS) after 5 treatments as compared to baseline.

SECONDARY OUTCOMES:
Change in gait parameters from baseline to 3 months post-treatment | Up to 3 months after last treatment session
  Change in walking up to 3 months after 5 treatments as compared to baseline as measured using a gait analysis system
Change in walking performance from baseline to 3 months post-treatment | Up to 3 months after last treatment session
  Change in walking performance up to 3 months after 5 treatments as compared to baseline as measured using the 10-meter walk test
Change in functional performance from baseline to 3 months post-treatment | Up to 3 months after last treatment session
  Change in functional performance up to 3 months after 5 treatments as compared to baseline as measured using the Fugl Meyer assessment
Change in muscle reaction from baseline to 3 months post-treatment | Up to 3 months after last treatment session
  Change in muscle reaction up to 3 months after 5 treatments as compared to baseline as measured using the H-reflex
Change in subject's self-assessment of their spasticity from baseline to 3 months post-treatment | Up to 3 months after last treatment session
  Change in subject's self-assessment of their spasticity up to 3 months after 5 treatments as compared to baseline as measured using an 11-point Numerical Rating Scale
Change in subject's quality of life from baseline to 3 months post-treatment | Up to 3 months after last treatment session
  Change in subject's self-assessment of quality of life up to 3 months after 5 treatments as compared to baseline as measured using the SF-36 scale

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Corvol, MD, PhD, Principal Investigator — Institut du Cerveau et de la Moelle épinière
Locations (1):
- Centre d'investigation clinique, Institut du Cerveau et de la Moelle, Paris, France

REFERENCES:
- [Background] Paget-Blanc A, Chang JL, Saul M, Lin R, Ahmed Z, Volpe BT. Non-invasive treatment of patients with upper extremity spasticity following stroke using paired trans-spinal and peripheral direct current stimulation. Bioelectron Med. 2019 Jul 23;5:11. doi: 10.1186/s42234-019-0028-9. eCollection 2019. PMID 32232101